CLINICAL TRIAL: NCT02133963
Title: Sleep Dysregulation and Neuroendocrine Stress Reactivity: Towards a Biopsychosocial Model of Vulnerability to Postpartum Depression
Brief Title: Determining Relationships Among Maternity Stress & Sleep
Acronym: DREAMSS
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Principal Investigator, Shannon Crowley, PhD, Postdoctoral Fellow, University of North Carolina, Chapel Hill
Other Study IDs: 13-3229
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Postpartum Depression; Depression
Keywords: depression; postpartum depression; pregnancy; perinatal depression; sleep; life stress
MeSH Terms: conditions — Depression, Postpartum; Depression; Stress, Psychological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma, Adrenocorticotropic hormone (ACTH), Cortisol
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- women with no history of depression: Non-Probability Sample of women with no history of depression
- women with a past depression history: Non-Probability Sample of women with a past history of depression

SUMMARY:
Psychosocial factors, including a previous history of depression, recent stressful life events, sleep disturbances during pregnancy, and depression and/or anxiety during pregnancy have been shown to be associated with an increased risk for the development of postpartum depression (PPD). Biological mechanisms underlying the relationships among these psychosocial risk factors for PPD, and the development of PPD, remain unclear. However, evidence from non-perinatal populations suggest that dysregulation in stress-reactive neuroendocrine factors may play a role. The primary objectives of this study are: (1) to assess the feasibility of enrolling second trimester pregnant women, with or without depression histories, into a laboratory-based study protocol which includes a mild psychosocial stressor and the collection of venous blood for the measurement of stress-reactive adrenocorticotropic hormone (ACTH) and cortisol; (2) to assess the feasibility of retaining participants, for a brief postpartum phone interview, after completion of the second trimester assessments; and (3) to establish proof of concept for measuring group differences, between women with or without depression histories, in second trimester prenatal measures of neuroendocrine stress reactivity, depressive and anxious symptoms, recent stressful life events, and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women in their 2nd trimester of a singleton pregnancy
* women between 18-45 years of age
* women with a past history of depression
* women with no past history of depression

Exclusion Criteria:

* under 18 years of age
* over 45 years of age
* pregnancy gestation > 22 weeks at study enrollment
* multiparity
* non-singleton pregnancy
* prior termination of pregnancy at >12 weeks gestation
* prior loss of pregnancy >2 times at <12 weeks gestation
* prior history of stillbirth
* current substance use (alcohol and/or elicit drugs)
* current chronic steroid use
* current use of antidepressants, anti-anxiety medications, mood-stabilizers, psychotropic medications, progesterone treatment, or sleep medications
* current tobacco use
* diagnosed obstructive sleep apnea,
* diagnosed restless legs syndrome (RLS)
* certain cancers
* pre-gestational diabetes
* a body mass index (BMI) of > 40kg/m2 just prior to pregnancy
* chronic hypertension (documented or taking medication for hypertension)
* gestational hypertension
* preeclampsia
* current anemia
* current or past history of psychosis, schizoaffective disorder,or bipolar disorder
* current depression

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample of pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of the study protocol during the prenatal phase. Feasibility will be defined by the successful completion of enrollment and stress testing lab visits in 13 out of the 15 participants designed per group. | 20-22 weeks gestation through 22-24 weeks gestation

SECONDARY OUTCOMES:
Feasibility with respect to the ability to retain participants / avoid attrition, which will be defined as having at least 90% of participants who completed the prenatal phase of the study, also complete one of the postpartum phone interviews. | Phone interviews will be administered at 8 weeks and 12 weeks postpartum.
The investigators will test for group differences, between women with or without depression histories, in stress reactivity of cortisol [calculated using area under the curve (AUC)] to a mild psychosocial stressor paradigm. | The mild psychosocial stressor paradigm will occur during the stress testing lab visit, which will be scheduled during gestational weeks 22-24
  The investigators will use a two-group t-test, or a Mann-Whitney-Wilcoxon test for non-normal distributions, to test for group differences in stress reactivity of cortisol [calculated using area under the curve (AUC)] to a mild psychosocial stressor paradigm.
The investigators will test for group differences, between women with or without depression histories, in stress reactivity of adrenocorticotropic hormone ACTH [calculated using area under the curve (AUC)] to a mild psychosocial stressor paradigm. | The mild psychosocial stressor paradigm will occur during the stress testing lab visit, which will be scheduled during gestational weeks 22-24
  The investigators will use a two-group t-test, or a Mann-Whitney-Wilcoxon test for non-normal distributions, to test for group differences in stress reactivity of adrenocorticotropic hormone (ACTH) [calculated using area under the curve (AUC)] to a mild psychosocial stressor paradigm.
The investigators will use a two-group t-test, or a Mann-Whitney-Wilcoxon test for non-normal distributions, to test for group differences in prenatal depressive symptoms using the Endinburgh Postnatal Depression Scale (EPDS). | The Endinburgh Postnatal Depression Scale (EPDS) will be administered during the enrollment visit, scheduled during gestational weeks 20-22.
The investigators will use a two-group t-test, or a Mann-Whitney-Wilcoxon test for non-normal distributions, to test for group differences in prenatal anxious symptoms using the Spielberger State-Trait Anxiety Inventory (STAI), trait version. | The trait version of the Spielberger State-Trait Anxiety Inventory (STAI) will be administered during the enrollment visit, scheduled during gestational weeks 20-22.
The investigators will use a two-group t-test, or a Mann-Whitney-Wilcoxon test for non-normal distributions, to test for group differences in recent stressful life events (last 6 months) using the Life Events Scale (LES). | The Life Events Scale (LES) will be administered during the enrollment visit, scheduled during gestational weeks 20-22.
The investigators will use a two-group t-test, or a Mann-Whitney-Wilcoxon test for non-normal distributions, to test for group differences in prenatal sleep quality (past 30 days) using the Pittsburgh Sleep Quality Index (PSQI). | The Pittsburgh Sleep Quality Index (PSQI) will be administered during the enrollment visit, scheduled during gestational weeks 20-22.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon K Crowley, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Susan S Girdler, PhD, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States